CLINICAL TRIAL: NCT06860724
Title: Linking Affective Dynamics in Response to Daily Stress to Peripheral Vascular Function in Working Age Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2270844; P20GM113125 (NIH)
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: stress; affect; endothelial function
MeSH Terms: conditions — Depressive Disorder, Major | interventions — NG-Nitroarginine Methyl Ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy adults (Active Comparator): non-depressed healthy adults
  Interventions: Other: NG-nitro-L-arginine methyl ester (L-NAME)
- adults with major depressive disorder (Experimental): adults with major depressive disorder (unmedicated)
  Interventions: Other: NG-nitro-L-arginine methyl ester (L-NAME)

INTERVENTIONS:
Other: NG-nitro-L-arginine methyl ester (L-NAME) — Acute local perfusion of L-NAME (15 mM) directly to the microvasculature will be used to inhibit NO synthase.

SUMMARY:
The objective of this proposal is to determine whether heightened negative affective responsivity (NA-R) to daily stressors is related to blunted nitric oxide (NO)-mediated endothelium-dependent dilation (EDD) in working age adults and the extent to which this association is impacted by major depressive disorder (MDD).

DETAILED DESCRIPTION:
Convincing evidence indicates that the deleterious impacts of psychosocial stress on emotional well-being and behavioral health are likely major contributors to excessive cardiovascular disease (CVD) risk in middle-aged and younger adults. In line with this, heightened negative affective (i.e., emotional) responsivity (NA-R) to daily stressors predicts CVD morbidity and mortality. Importantly, NA-R to daily stressors-the naturally occurring but unexpected hassles and challenges that arise out of routine everyday life (e.g., argument with a partner, pressing work deadline)-is most pronounced in 'working age adults' (18-55 yrs). Unfortunately, these effects appear further compounded in adults with major depressive disorder (MDD), an increasingly prevalent mood disorder whose core pathology is characterized by dysregulated affective dynamics. However, the physiological mechanisms linking dysregulated daily stress-related affective dynamics to poorer long-term cardiovascular health trajectories in working age adults remain incompletely understood. Our global hypothesis that affective dysregulation in response to daily stressors contributes to worsening endothelial health in working age adults, the effects of which are exacerbated in adults with MDD. Working age non-depressed healthy adults (HA) and adults with MDD (unmedicated) will participate. Multiple dynamic aspects of affective regulation and daily stress processes will be assessed during routine everyday life for 14 consecutive days (mobile app). On the days immediately before and after these ambulatory assessments, the mechanistic regulation of microvascular endothelial function will be assessed (in vivo; physiological and pharmacological approaches).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-55 yrs
* Non-depressed health adults (HA) will have no evidence of current or lifetime history of major psychiatric illness, assessed by the MINI and self-report and confirmed by a Licensed Clinical Psychologist
* Adults with major depressive disorder (MDD) must meet the DSM-5 criteria for MDD and be currently symptomatic, assessed by the MINI and confirmed by a Licensed Clinical Psychologist; participants with co-morbid anxiety, stress, and trauma-related disorders will be included
* Absence of unstable or chronic clinical disease, including cardiovascular, metabolic, renal, hepatic, autonomic, autoimmune, or dermatological disease, as determined by medical history, physical examination, blood chemistries, and 12-lead resting electrocardiogram; however, to ensure a more generalizable sample, adults with elevated systolic BP (<130mmHg), direct low-density lipoprotein (<160mg/dl), and glucose (HbA1c <5.7%) will be included
* Participants must have a level of understanding of the English language sufficient to provide informed consent and to agree to all tests and procedures, as well as the capacity and willingness to attend all study related visits and to comply with the study protocol

Exclusion Criteria:

Subjects will be excluded at the discretion of the PI/collaborating clinicians or for any of the following reasons:

* <18 or >55 yrs
* Lifetime or current co-morbid neuropsychiatric disease (bipolar disorder, psychotic disorders, schizophrenia, eating disorders, obsessive-compulsive disorder, alcohol or substance use disorders)
* Serious and imminent active suicidal/homicidal ideation with intent, plans, or behaviors, determined by the Licensed Clinical Psychologist or other clinical study team staff
* Diagnosed chronic clinical disease, including cardiovascular, metabolic, renal, hepatic, autonomic, autoimmune, or dermatological disease, as determined by medical history, physical examination (resting systolic BP ≥130mmHg, body mass index ≥35 kg/m2), clinically significant abnormal blood chemistries (direct low-density lipoprotein ≥160mg/dl, HbA1c≥5.7%), and clinically significant abnormal 12-lead resting ECG
* Current or recent use (within last 8 wks) of medications that alter cardiovascular function or psychoactive or psychopharmacological drugs [including (but not limited to) antidepressants, antipsychotics, benzodiazepines, mood stabilizers, sedatives/hypnotics, dopaminergic agents, stimulants, buspirone, and triptans]
* Tobacco use (including electronic cigarettes)
* Females who are pregnant, breastfeeding, or planning to become pregnant; female subjects of child-bearing age must have a negative urine pregnancy test on the day of all experimental visits
* Current or past use of hormone replacement therapy
* Allergy to study drugs or pharmacological agents

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Nitric oxide (NO)-mediated endothelium-dependent dilation (EDD) | immediately before and after the 14-day testing cycle
  A standard local heating protocol will be used to elicit EDD and the NO-dependent portion of this response will be determined pharmacologically (local perfusion of L-NAME). Vascular conductance will be calculated (CVC=flux/mean arterial pressure) and normalized to the site-specific maximum. NO-mediated EDD will be calculated as the percent change from the local heating-induced plateau to the post-L-NAME plateau.
Negative affective responsivity (NA-R) to daily stressors | immediately after the 14-day testing cycle
  NA-R to daily stressors will be operationalized as the within-person slope of the change in negative affect on stressor days compared to stressor-free days and calculated using multilevel modeling. The models for computing NA-R slopes will use maximum likelihood estimation (MLE), which accounts for participants potentially providing different numbers of diary days, and will include stressor exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No